CLINICAL TRIAL: NCT04434651
Title: Effect of Sphenopalatine Ganglion Block on Intracranial Pressure and Cerebral Venous Outflow Oxygenation During Craniotomy for Supratentorial Brain Tumors.
Brief Title: Effect of SPGB on ICP and Oxygenation of Cerebral Venous Outflow in Craniotomy for Cerebral Tumors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, Lecturer, Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6180
Record Dates: First submitted 2020-06-13; First posted 2020-06-17 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Tumor
Keywords: SPGB; ICP; CBF; AVDO2
MeSH Terms: interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: This study will be performed in the Neurosurgical operating room and included 52 patients allocated into two groups: the treatment group (block group) and the control group (non-block group). 26 patients enrolled in block group and 26 patients in non-block group.
  Intraoperative ICP monitoring by subdural ICP monitors will be done every 20 minutes in both block and non- block group.
  Jugular venous bulb oxygen saturation changes will be recorded every 20 minutes in block and non- block.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Block group (A) (Experimental): 26 patients who will be subjected to a neurosurgical intervention for removal of supratentorial brain tumor. Supratentorial brain tumors with shift of the mid-line <10 mm evaluated by CT scan [computerized tomography] . SPGB will be performed using 2 % lidocaine before induction of anesthesia.
  The anesthesia induced by IV anesthetics and maintained by Isoflurane. ICP, Jugular venous bulb oxygen saturation, and AVDO2 will be assessed every 20 minutes.
  Interventions: Procedure: SPGB
- control sham group (B) (Sham Comparator): 26 patients who will be subjected to a neurosurgical intervention for removal of supratentorial brain tumor. Supratentorial brain tumors with shift of the mid-line <10 mm evaluated by CT scan [computerized tomography] . SPGB will be performed using normal saline.The anesthesia induced by IV anesthetics and maintained by Isoflurane. ICP, Jugular venous bulb oxygen saturation, and AVDO2 will be assessed every 20 minutes
  Interventions: Procedure: SPGB

INTERVENTIONS:
Procedure: SPGB — Sphenopalatine Ganglion Block using 2% lidocaine in block group. Sphenopalatine Ganglion Block is performed by a hollow culture swab that is connected with a 21-gauge a syringe filled with three ml 2% lidocaine, inserted parallel to the floor of the nose until resistance is felt. The swab is at the posterior pharyngeal wall superior to the middle turbinate. The applicator was kept in the nostril for five to ten mins. The same procedure is done also in the second nostril SPGB using normal saline is performed in the control group
  Other Names: Sphenopalatine ganglion block

SUMMARY:
This study aims to investigate the effect of Sphenopalatine Ganglion Block on ICP and arterio- jugular venous oxygen difference (AJVDO2) and jugular bulb oxygen saturation (SjVO2). Throughout this study, the efficacy of Sphenopalatine Ganglion Block as scalp block in craniotomy operation will be assessed, and the effect of SPGB on cerebral hemostasis during craniotomy will be evaluated by monitoring of both ICP, AJVDO2 and SjVO2.

DETAILED DESCRIPTION:
This study was performed in the Neurosurgical operating room and included 52 patients allocated into two groups: the treatment group (block group) and the control group (non-block group). 26 patients enrolled in block group and 26 patients in non-block group.

Intraoperative ICP monitoring by subdural ICP monitors will be done every 20 minutes in both block and non- block groups until craniotomy has been occurred, then at the time of closure of the dura . Arterio- jugular venous oxygen difference and Jugular venous bulb oxygen saturation changes will be recorded every 20 minutes in block and non- block groups throughout time of the surgery till closure of the dura.

ELIGIBILITY:
Inclusion Criteria:

* Patients who prepared for a neurosurgical intervention for elective supratentorial tumor removal
* ASA 1 and 2
* Age above 18 years and below 65 years
* Fully conscious patients.

Exclusion Criteria:

* Patients with cardiovascular and respiratory diseases
* Pregnancy
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Intracranial Pressure | Every 20 minutes until time of initial craniotomy, then again after the dura was sutured.
  ICP changes checked by a subdural ICP monitor that positioned after the first burr hole at the opposite side of the tumor immediately after induction of anesthesia. ICP monitoring will be conducted every 20 minutes until time of initial craniotomy and at time of closure of the dura.

SECONDARY OUTCOMES:
Jugular venous bulb oxygen saturation and cerebral arteriovenous oxygen content difference. | Every 20 minutes throughout the operation period.
  Jugular venous bulb oxygen saturation will be measured then AVDO2 will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa Abdelhaleem, MD, Principal Investigator — Faculty of Medicine, Zagazig University, Zagazig, Egypt.
Locations (1):
- Faculty of Medicine, Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
it will be available after completion of study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available 3 months after publication of study
Access Criteria: By contacting the principal investigator
URL: https://register.clinicaltrials.gov/prs/app

REFERENCES:
- [Background] Kaye A, Kucera IJ, Heavner J, Gelb A, Anwar M, Duban M, Arif AS, Craen R, Chang CT, Trillo R, Hoffman M. The comparative effects of desflurane and isoflurane on lumbar cerebrospinal fluid pressure in patients undergoing craniotomy for supratentorial tumors. Anesth Analg. 2004 Apr;98(4):1127-1132. doi: 10.1213/01.ANE.0000105862.78906.3D. PMID 15041612
- [Background] Feldman Z, Robertson CS. Monitoring of cerebral hemodynamics with jugular bulb catheters. Crit Care Clin. 1997 Jan;13(1):51-77. doi: 10.1016/s0749-0704(05)70296-7. PMID 9012576